CLINICAL TRIAL: NCT03720782
Title: Multi-center Study of the Safety and Performance of Primary Total Knee Arthroplasty With LEGION™ Porous HA Tibial Baseplates (With and Without Holes) and/or the LEGION™ Porous HA CR Femoral Component in US Centers
Brief Title: Safety and Performance Study of the Legion Porous System in Total Knee Arthroplasty
Status: Active, not recruiting | Type: Observational
Sponsor: Smith & Nephew, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: LEGHA.PMCF.2018.07
Record Dates: First submitted 2018-10-19; First posted 2018-10-25 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-04

CONDITIONS: Total Knee Arthroplasty
Keywords: Legion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

INTERVENTIONS:
Device: LEGION Porous HA Tibial Baseplate and/or the LEGION Porous HA CR Femoral Component — LEGION Porous HA Tibial Baseplate (with and without holes) and/or the LEGION Porous HA CR Femoral Component

SUMMARY:
The purpose of this research is to collect data on patients that had the Legion Porous HA Tibial Baseplates and/or the Legion Porous HA Femoral component implanted in the past. Smith & Nephew will evaluate the safety and performance of these implants for 10 years post-surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Subject received primary TKA with the LEGION Porous HA Tibial Baseplates (either with holes or without holes) and/or the LEGION Porous HA CR Femoral Component, due to degenerative joint disease (primary diagnosis of osteoarthritis, post-traumatic arthritis, or degenerative arthritis).
2. Subject received primary TKA between 24 and 60 months prior to the time of consent.

   Inclusion criteria for prospective follow-up (subjects must meet criteria 1 & 2 from above and criteria 3,4 and 5 below):
3. Subject agrees to consent and to follow the prospective study visit schedule (as defined in the study protocol and informed consent form) by signing the IRB/IEC approved informed consent form.
4. Subject must be available through ten (10) years postoperative follow-up.
5. Subject is able to read, understand, and communicate responses to Patient Reported Outcome assessments in English.

Exclusion Criteria:

Exclusion criteria for retrospective chart review - Any one (1) of the following criteria will disqualify a potential subject from participation in the retrospective chart review:

1. Subject received TKA on the contralateral knee as a revision for a previously failed total or unicondylar knee arthroplasty
2. Subject has ipsilateral hip arthritis resulting in flexion contracture.
3. At the time of enrollment, subject has one or more of the following arthroplasties that are not fully healed and well-functioning, as determined by the investigator: Ipsilateral or contralateral primary total hip arthroplasty or hip resurfacing arthroplasty; Contralateral primary total knee or unicondylar knee arthroplasty.
4. Subject has a condition that may interfere with the TKA survival or outcome (e.g. Paget's or Charcot's disease, vascular insufficiency, lupus, muscular atrophy, uncontrolled diabetes, moderate to severe renal insufficiency or neuromuscular disease).
5. Subject has a known allergy to one or more of its components of the study device.
6. Subject is entered in another drug, biologic, or device study or has been treated with an investigational product in the past 30 days.

   Exclusion criteria for prospective follow-up - Any one (1) of the criteria from 1-6 above will disqualify a potential subject from participation in the prospective follow-up) as will any one (1) of the below criteria 7, 8 and 9:
7. Subject, in the opinion of the Principal Investigator (PI), has an emotional or neurological condition that would pre-empt their ability or willingness to participate in the study including mental illness, mental retardation, drug or alcohol abuse.
8. Subject is known to be at risk for loss to follow-up, or failure to return for scheduled visits.
9. Subject is found to have had a revision of the study device(s).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Maximum of 150 subjects enrolled to obtain a minimum of 150 implanted components:
  * Maximum of 75 subjects to obtain a minimum of 75 implanted tibial baseplate components (with or without holes) to attain 30 evaluable baseplates with holes and 30 evaluable baseplates without holes (i.e. a combined total of 60 evaluable implanted baseplate components)
  * Maximum of 75 subjects to obtain a minimum of 75 implanted LEGION Porous HA CR Femoral Components to attain 60 evaluable components.
  Note: Some subjects may have received both the LEGION Porous HA Tibial Baseplate (with or without holes) and the LEGION Porous HA CR Femoral Component during their TKA procedure.
Sampling Method: Non-Probability Sample
Enrollment: 118 (Actual)
Dates: Start 2019-05-22 (Actual); Primary Completion 2031-01-23 (Estimated); Study Completion 2032-12-31 (Estimated)

PRIMARY OUTCOMES:
Implant survivorship 10 years post-surgery | 10 years

SECONDARY OUTCOMES:
Quality of life - KOOS JR | 10 years
  Patient Reported Outcomes using Knee Injury and Osteoarthritic Outcome Scores (KOOS JR) questionnaire
Quality of Life - Forgotten Joint Score (FJS) | 10 years
  Patient Reported Outcomes using Forgotten Joint Score (FJS) questionnaire
Quality of life - EQ-5D-5L | 10 years
  Patient Reported Outcomes using EuroQol Five Dimensions Questionnaire (EQ-5D - 3L) questionnaire
Implant survivorship | 5 years
  Implant Survivorship at 5 years defined as the cumulative proportion of knee-implanted components without a revision
Radiographic findings | 10 years
  X-ray of implanted knee- 3 views (AP, Lateral and Skyline/Merchant) to observe any radiographic findings that may include; Heterotopic ossification, oteolysis, femoral notching, evidence of poly wear, radiolucencies.

CONTACTS AND LOCATIONS:
Overall Officials: Karlie Morgan, Study Chair — Smith & Nephew, Inc.
Locations (2):
- United States (2):
  - Twin Cities Orthopedics, Coon Rapids, Minnesota
  - Saint Louis University Hospital, Dept. of Orthopaedic Surgery, St Louis, Missouri